CLINICAL TRIAL: NCT00600925
Title: A Randomized, Controlled, Phase 3 Study of Gentamicin-Collagen Sponge in General Surgical Subjects at Higher Risk for Surgical Wound Infection
Brief Title: A Study of an Antibiotic Implant in General Surgical Subjects at Higher Risk for Surgical Wound Infection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Innocoll (Industry)
Collaborators: Duke University (Other); Premier Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: INN-SWI-002; NCT01150773 (obsolete NCT alias)
Record Dates: First submitted 2008-01-14; First posted 2008-01-25 (Estimated); Results first posted 2021-09-24 (Actual); Last update posted 2021-09-24 (Actual); Status verified 2021-09

CONDITIONS: Colorectal Surgery; Surgical Wound Infection
Keywords: Colorectal surgery
MeSH Terms: conditions — Surgical Wound Infection | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Insertion of 2 gentamicin-collagen sponges before closure of the laparotomy (each 10 x 10 cm sponge contains 280 mg collagen and 130 mg gentamicin).
  Interventions: Drug: gentamicin-collagen sponge dipped in saline
- 2 (No Intervention): Standard of care, ie, no gentamicin-collagen sponge.

INTERVENTIONS:
Drug: gentamicin-collagen sponge dipped in saline — 2 gentamicin-collagen sponges inserted before closure of the laparotomy
  Arms: 1

SUMMARY:
The purpose of this study is to determine whether the gentamicin-collagen sponge is safe and effective for preventing surgical wound infections in patients undergoing colorectal surgery.

DETAILED DESCRIPTION:
Surgical wound infection (SWI) is a significant problem in colorectal surgery. Despite the use of routine bowel preparation and prophylactic antibiotics the incidence of SWI is at least 15% in patients undergoing colorectal surgical procedures.Therefore, there is a long unmet need for an intervention that can reduce the incidence and severity of SWIs in patients undergoing colorectal surgery.

Gentamicin is an antibiotic that is effective in treating certain kinds of infection. Collagen is a protein that is found in all mammals. The gentamicin-collagen sponge is a thin flat sponge made out of collagen that comes from cow tendons and containing gentamicin. When inserted into a surgical site, the collagen breaks down and the gentamicin is released at the site but very little is absorbed into the blood stream. The high levels of antibiotic at the surgical site may prevent an infection at the surgical site.

Outside of the United States more than 3,500 subjects have received treatment in clinical studies with the gentamicin-collagen sponge, primarily for orthopedic, intraabdominal, and cardiothoracic surgeries or wound infections following surgical procedures or traumatic events.

In this study, all subjects will be given treatment that is normally given to prevent surgical infections. For subjects randomly assigned to the gentamicin-collagen sponge treatment group, 2 sponges will be inserted into the surgical wound immediately before the surgeon closes it. The control group will receive no collagen sponge.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to undergo nonemergent colon and/or rectal surgical procedures involving a laparotomy incision of at least 7 cm in length or greater. List of eligible procedures: Left Hemicolectomy, Transverse Colectomy, Segmental/Sleeve Left Colon Resection, Total Abdominal Colectomy With Ileorectal Anastomosis, Total Abdominal Colectomy With Ileostomy, Total Abdominal Proctocolectomy (Portion Of Specimen To Be Extracted Via Laparotomy), Low Anterior Resection, Sigmoid Resection, Non-Emergent Hartmann's Procedure, Colotomy With Polypectomy Distal To Hepatic Flexure, Colostomy Takedown Through Laparotomy (Not Peristomal) Incision, Ileo-Pouch Anal Anastomosis, Abdominal Perineal Resection of the Rectum
* Have the capacity to understand and sign an informed consent form.
* Are male or female and > 18 years of age.
* If female, be postmenopausal (no menstrual period for a minimum of 1 year), or surgically sterilized (does not have a uterus or has had bilateral tubal ligation). Females of child-bearing potential must have a negative serum pregnancy test on entry in the study, and agree to use adequate birth control during the study and for 60 days after the administration of study agent.
* Agree to be available for evaluation from baseline until final evaluation at 60 days postsurgery.

Exclusion Criteria:

* Known history of hypersensitivity to gentamicin or bovine collagen.
* Undergoing emergency surgery (urgent surgery is allowed if informed consent is obtained and the study procedures can be performed). Emergency surgery includes cases where standard bowel preparation and other preoperative assessments cannot be done.
* Undergoing a significant concomitant surgical procedure (e.g., hysterectomy). The following concomitant procedures are allowed: appendectomy, cholecystectomy, oophorectomy, liver biopsy/wedge resection (but not liver resection).
* Undergoing a laparoscopic, laparoscopic-assisted, or other minimally invasive surgical approach involving a laparotomy incision less than 7 cm.
* History of prior laparotomy within the last 60 days of this planned procedure.
* Planned to undergo a second laparotomy or colorectal surgical procedure (e.g. colostomy or ileostomy takedown) within 60 days of this planned first procedure.
* Evidence preoperatively of any of the following: sepsis, severe sepsis, or septic shock (note that SIRS alone is not an exclusion criterion)
* Current abdominal wall infection/surgical site infection from previous laparotomy/laparoscopy or for any reason.
* Receiving antibiotic therapy within the 1 week prior to the date of surgery.
* Preoperative evaluation suggests intra-abdominal process that might preclude full closure of the skin.
* History of ongoing treatment (e.g. chemotherapy, radiation) for non-colorectal cancer.
* Recent history of significant drug or alcohol abuse.
* Preoperative prothrombin time (PT) > 1.5 times upper limit of normal
* Pregnant, lactating, or of childbearing potential not practicing a birth control method with a high degree of reliability
* Postsurgical life expectancy ≤ 60 days, in the investigator's or sponsor's opinion.
* Refusal to accept medically indicated blood products.
* Previous participation in this or any other active Innocoll Gentamicin-Collagen Sponge study.
* Participation within 30 days before the start of this study in any experimental drug or device study, or currently participating in a study in which the administration of investigational drug or device within 60 days is anticipated.
* Surgeon does not believe that it will be possible to insert 2 sponges above the fascia in the patient (e.g. in a very thin patient planned to have a small incision)
* Patients with anterior abdominal wall mesh that is not planned to be completely removed during the planned procedure.
* Presence of prosthetic cardiac valve.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 602 (Actual)
Dates: Start 2008-01; Primary Completion 2009-03 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Prior, Study Director — Innocoll
Locations (39):
- United States (39):
  - Florence, Alabama
  - Mobile, Alabama
  - Laguna Hills, California
  - Los Angeles, California
  - Stanford, California
  - Aurora, Colorado
  - Denver, Colorado
  - Tampa, Florida
  - Weston, Florida
  - Atlanta, Georgia
  - Indianapolis, Indiana
  - Louisville, Kentucky
  - New Orleans, Louisiana
  - Baltimore, Maryland
  - Detroit, Michigan
  - Duluth, Minnesota
  - Minneapolis, Minnesota
  - St Louis, Missouri
  - Albany, New York
  - Brooklyn, New York
  - New York, New York
  - Syracuse, New York
  - Chapel Hill, North Carolina
  - Durham, North Carolina
  - Greensboro, North Carolina
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Columbus, Ohio
  - Oklahoma City, Oklahoma
  - Portland, Oregon
  - Hershey, Pennsylvania
  - Philadelphia, Pennsylvania
  - Nashville, Tennessee
  - Dallas, Texas
  - Houston, Texas
  - Temple, Texas
  - Burlington, Vermont
  - Seattle, Washington
  - Tacoma, Washington

REFERENCES:
- [Derived] Bennett-Guerrero E, Pappas TN, Koltun WA, Fleshman JW, Lin M, Garg J, Mark DB, Marcet JE, Remzi FH, George VV, Newland K, Corey GR; SWIPE 2 Trial Group. Gentamicin-collagen sponge for infection prophylaxis in colorectal surgery. N Engl J Med. 2010 Sep 9;363(11):1038-49. doi: 10.1056/NEJMoa1000837. Epub 2010 Aug 4. PMID 20825316

RESULTS

PARTICIPANT FLOW:
Groups:
- Gentamicin Group: Insertion of 2 gentamicin-collagen sponges before closure of the laparotomy (each 10 x 10 cm sponge contains 280 mg collagen and 130 mg gentamicin).
  gentamicin-collagen sponge dipped in saline: 2 gentamicin-collagen sponges inserted before closure of the laparotomy
- Control: Standard of care, ie, no gentamicin-collagen sponge.
Period: Overall Study
Arm/Group | Gentamicin Group | Control
Started | 300 | 302
Completed | 300 | 302
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Gentamicin Group Group: Insertion of 2 gentamicin-collagen sponges before closure of the laparotomy (each 10 x 10 cm sponge contains 280 mg collagen and 130 mg gentamicin).
  gentamicin-collagen sponge dipped in saline: 2 gentamicin-collagen sponges inserted before closure of the laparotomy
- Control Group: Standard of care, ie, no gentamicin-collagen sponge.
- Total: Total of all reporting groups
Arm/Group | Gentamicin Group Group | Control Group | Total
Number analyzed (Participants) | 300 | 302 | 602
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.9 (15.36) | 56.5 (15.81) | 56.7 (15.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 181 | 158 | 339
  Male | 119 | 144 | 263
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 6 | 8
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 2
  Black or African American | 22 | 19 | 41
  White | 272 | 273 | 545
  More than one race | 2 | 4 | 6
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Surgical Wound Infections From Surgery Through Post-operative Day 60
Description: Primarily, efficacy will be evaluated by a comparison between the 2 study groups of the incidence of surgical wound infections (involving the laparotomy incision) that occur within the period from surgery through postop day 60.
Time Frame: assessed at Postop Day 1, 2, 3, 7, 30 & 60
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | Gentamicin Group | Control
Number analyzed (Participants) | 300 | 302
Participants | 90 | 63

2. Secondary Outcome: Number of Participants Who Had Superficial Incisional Surgical Wound Infection
Description: Number of Participants who had superficial incisional surgical wound infection, based on CDC criteria adjudicated by an independent blinded committee
Time Frame: assessed at Postop Day 1, 2, 3, 7, 30 & 60
Measure: Count of Participants; unit: Participants
Arm/Group | Gentamicin Group | Control
Number analyzed (Participants) | 300 | 302
Participants | 61 | 41

3. Secondary Outcome: The Effect of the Gentamicin-collagen Sponge on the Proportion of Patients With Deep Incisional Surgical Wound Infection
Description: The proportion of subjects who had deep incisional SWI, based on Centers for Disease Control and Prevention (CDC) criteria adjudicated by an independent blinded committee
Time Frame: assessed at Postop Day 1, 2, 3, 7, 30 & 60
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | Gentamicin Group | Control
Number analyzed (Participants) | 300 | 302
Participants | 25 | 18

4. Secondary Outcome: The Effect of the Gentamicin-collagen Sponge on the ASEPSIS Score
Description: Mean (SD) ASEPSIS Score Through 60 Days Postoperatively - brief assessment of surgical wound on post-operative Days 3, 4, 5, 6, and 7 (or discharge if earlier) and then questionnaire/phone call on post-operative Days 30 and 60. Score from each time point is added up and the mean score is reported. Used to compare antibiotic regimens for their effectiveness in preventing or treating wound sepsis, well-defined criteria for outcome are needed. A method of assessing wound healing has been devised that defines carefully the characteristics to be considered and how they are to be awarded points. Objective criteria are also included in the assessment. Points are given for the need for Additional treatment, the presence of Serous discharge, Erythema, Purulent exudate, and Separation of the deep tissues, the Isolation of bacteria, and the duration of inpatient Stay (ASEPSIS). The higher the points the worse outcome. Maximum Points would be 60. Minimum points would be 0
Time Frame: Days 3, 4, 5, 6, and 7 (or discharge if earlier) and then questionnaire/phone call on post-operative Days 30 and 60.
Population: ITT population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Gentamicin Group | Control
Number analyzed (Participants) | 299 | 299
score on a scale | 6.1 (10.38) | 5.2 (10.99)

5. Secondary Outcome: The Effect of the Gentamicin-collagen Sponge on Length of Hospital Stay Postoperatively.
Time Frame: Immediate post operative period
Population: ITT population
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Gentamicin Group | Control
Number analyzed (Participants) | 300 | 302
days | 7.5 (6.19) | 7.3 (5.42)

6. Secondary Outcome: Number of Participants Who Were Rehospitalized for Surgical Wound Infection Within 60 Days Post-operatively
Description: The effect of the gentamicin-collagen sponge on rehospitalization for surgical wound infection.
Time Frame: Through 60 days after surgery
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | Gentamicin Group | Control
Number analyzed (Participants) | 300 | 302
Participants | 21 | 13

ADVERSE EVENTS:
Time Frame: Subjects remained enrolled into the study until 60 days post-operatively
Description: The ITT population is analyzed as randomized, while the safety population is analyzed as treated. There were 4 patients who were randomized to the gentamicin group who were not treated with the sponge. The analyses based on the safety population includes the 302 patients randomized to placebo plus these additional 4 patients.
Arm/Group | Gentamicin Group Group | Control Group
All-Cause Mortality (participants affected / at risk) | 1/296 | 5/306
Serious Adverse Events (participants affected / at risk) | 114/296 | 101/306
Other Adverse Events (participants affected / at risk) | 294/296 | 302/306
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gentamicin Group Group (N=296) | Control Group (N=306)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Pernicious anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Splenic infarcation (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 2 (2)
Atrial Fibrillation (Cardiac disorders) | 3 (3) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 2 (2)
Colonic fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Crohn's disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Duodenal ulcer perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enterocutaneous fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Faecal volume increased (Gastrointestinal disorders) | 1 (1) | 2 (2)
Faecaloma (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric hypomotility (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastrointestinal hypomotility (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal motility disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inguinal hernia strangulated (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intra-abdominal haematoma (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 1 (1) | 2 (2)
Large intestine perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mesenteric panniculitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Peritonitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Proctalgia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 4 (4) | 0 (0)
Reflux oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 8 (8) | 10 (10)
Vomiting (Gastrointestinal disorders) | 3 (3) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Hepatobiliary disorders (General disorders) | 6 (6) | 1 (1)
Cholecystitis (General disorders) | 1 (1) | 1 (1)
Cholecystitis acute (General disorders) | 3 (3) | 0 (0)
Portal vein thrombosis (General disorders) | 2 (2) | 0 (0)
abdominal abcess (Infections and infestations) | 2 (2) | 3 (3)
Abdominal infection (Infections and infestations) | 1 (1) | 0 (0)
Abdominal sepsis (Infections and infestations) | 1 (1) | 1 (1)
Abdominal wall infection (Infections and infestations) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 0 (0) | 2 (2)
Catheter site infection (Infections and infestations) | 1 (1) | 0 (0)
Central line infection (Infections and infestations) | 1 (1) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1)
Emphysematous cholecystitis (Infections and infestations) | 1 (1) | 0 (0)
Endocarditis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Fungaemia (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Haematoma infection (Infections and infestations) | 1 (1) | 0 (0)
Pelvic abscess (Infections and infestations) | 9 (9) | 7 (7)
Pelvic infection (Infections and infestations) | 1 (1) | 0 (0)
Pelvic sepsis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2) | 2 (2)
Post procedural cellulitis (Infections and infestations) | 1 (1) | 1 (1)
Postoperative abscess (Infections and infestations) | 3 (3) | 1 (1)
Postoperative wound infection (Infections and infestations) | 19 (19) | 7 (7)
Rectal abscess (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 1 (1)
Soft tissue infection (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal infection (Infections and infestations) | 0 (0) | 1 (1)
Abdominal wound dehiscence (Injury, poisoning and procedural complications) | 7 (7) | 3 (3)
Anastomotic stenosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Deep vein thrombosis postoperative (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Gastrointestinal anastomotic leak (Injury, poisoning and procedural complications) | 8 (8) | 4 (4)
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 0 (0) | 4 (4)
Intestinal anastomosis complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Jaw fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural discharge (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Postoperative ileus (Injury, poisoning and procedural complications) | 30 (30) | 19 (19)
Postoperative wound complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Seroma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Therapeutic agent toxicity (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ulna fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ureteric injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Urethral injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Urinary retention postoperative (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound evisceration (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
wound secretion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
investigations (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Aspiration bronchial (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
international normalised ration decrease (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 14 (14) | 9 (9)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypovolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 4 (4) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Colon cancer metastatic (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hepatic neoplasm (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Metastatic neoplasm (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Nervous system disorders (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Cerebrovascular accident (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Paraplegia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Syncope (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Thalamic infarction (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Psychiatric disorders (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Confusional state (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Calculus ureteric (Renal and urinary disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal disorder (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 2 (2)
Renal failure acute (Renal and urinary disorders) | 3 (3) | 3 (3)
Renal failure chronic (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal infarct (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal tubular necrosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Female genital tract fistula (Reproductive system and breast disorders) | 1 (1) | 3 (3)
Pelvic haematoma (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 0 (0) | 1 (1)
Haemorrhage (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gentamicin Group Group (N=296) | Control Group (N=306)
Anaemia (Blood and lymphatic system disorders) | 70 (70) | 51 (51)
Leukocytosis (Blood and lymphatic system disorders) | 17 (17) | 14 (14)
Tachycardia (Cardiac disorders) | 46 (46) | 46 (46)
Abdominal Distension (Gastrointestinal disorders) | 70 (70) | 73 (73)
Abdominal pain (Gastrointestinal disorders) | 71 (71) | 81 (81)
Diarrhoea (Gastrointestinal disorders) | 23 (23) | 13 (13)
Nausea (Gastrointestinal disorders) | 167 (167) | 191 (191)
Vomiting (Gastrointestinal disorders) | 98 (98) | 79 (79)
Fatigue (General disorders) | 16 (16) | 16 (16)
Oedema Peripheral (General disorders) | 18 (18) | 21 (21)
Pyrexia (General disorders) | 57 (57) | 59 (59)
Post-operative Wound infection (Infections and infestations) | 47 (47) | 35 (35)
Urinary Tract Infection (Infections and infestations) | 22 (22) | 32 (32)
Abdominal Wound Dehiscence (Injury, poisoning and procedural complications) | 34 (34) | 17 (17)
Incision Site Pain (Injury, poisoning and procedural complications) | 119 (119) | 122 (122)
Post procedural Discharge (Injury, poisoning and procedural complications) | 57 (57) | 42 (42)
Post-operative Ileus (Injury, poisoning and procedural complications) | 23 (23) | 31 (31)
Post-operative Wound Complication (Injury, poisoning and procedural complications) | 33 (33) | 41 (41)
Procedural Pain (Injury, poisoning and procedural complications) | 81 (81) | 77 (77)
Blood Glucose Increased (Investigations) | 16 (16) | 18 (18)
Body Temperature Increased (Investigations) | 24 (24) | 21 (21)
Breath Sounds Abnorma (Investigations) | 26 (26) | 18 (18)
Urine Output Decreased (Investigations) | 25 (25) | 19 (19)
White Blood Cell Count Increased (Investigations) | 26 (26) | 18 (18)
Decreased Appetite (Metabolism and nutrition disorders) | 18 (18) | 18 (18)
Dehydration (Metabolism and nutrition disorders) | 16 (16) | 14 (14)
Hyperglycaemia (Metabolism and nutrition disorders) | 21 (21) | 20 (20)
Hypokalaemia (Metabolism and nutrition disorders) | 49 (49) | 45 (45)
Hypomagnesaemia (Metabolism and nutrition disorders) | 35 (35) | 28 (28)
Back Pain (Musculoskeletal and connective tissue disorders) | 15 (15) | 22 (22)
Dizziness (Nervous system disorders) | 33 (33) | 33 (33)
Headache (Nervous system disorders) | 16 (16) | 23 (23)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 15 (15) | 18 (18)
Pruritus (Skin and subcutaneous tissue disorders) | 22 (22) | 23 (23)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No